CLINICAL TRIAL: NCT06335628
Title: Volumetric Dimensional Changes After Surgical Pontic Site Development Procedures With Connective Tissue Graft or Collagen Matrix
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCT: CTG-VCMX
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Connective Tissue Graft; Volume Collagen Matrix Xenograft

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Connective Tissue Graft (CTG) (No Intervention): Volumetric changes between groups will be compared by matching intraoral scans before and after surgery (including follow-ups after 5 years) using the engineering software Geo-Magic®.
- Group B: Volume Collagen Matrix Xenograft (VCMX) Geistlich Fibro-Gide® (Experimental): The CTG (Group A) is the gold-standard for soft tissue augmentation, therefore it is considered the control group in this investigation.
  Interventions: Device: Geistlich Fibro-Gide®

INTERVENTIONS:
Device: Geistlich Fibro-Gide® — Geistlich Fibro-Gide® is intended to be used as an implantable device for regeneration and augmentation of soft tissue in oral and maxillofacial surgery.
  Arms: Group B: Volume Collagen Matrix Xenograft (VCMX) Geistlich Fibro-Gide®

SUMMARY:
The aim of this research project is to compare two surgical procedures to improve soft tissue volume. Both procedures have already been validated, but despite their great clinical relevance, little data exists in the literature. With this study, the investigators aim to evaluate volumetric changes of connective tissue graft versus biomaterial (membrane). In addition, further clinical measurements will be taken and patient satisfaction will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Age ≥ 18 years
* Willingness to sign informed consent and to participate in the study
* Single tooth gap or extended edentulous space in the lower or posterior jaw including a pontic site with a soft tissue deficiency.
* Tooth gap of ≥ 8 mm.
* Presence of natural or artificial opposing dentition
* Sufficient vertical interocclusal space of an implant restoration (7mm)
* Bounded by natural and periodontally stable teeth
* Treatment plan must include tooth replacement with an implant or tooth-supported fixed dental prosthesis.

Exclusion Criteria:

* Any physical or mental disorder that would interfere with the ability to perform adequate oral hygiene or the capability of providing written informed consent and compliance with the protocol
* Severe bruxism, clenching habits, or presence of oro-facial pain
* Uncontrolled diabetes mellitus (HbA1c >7.0)
* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.)
* Any active oral or systemic acute infections
* Currently receiving chemo- or radiotherapy or a history of radiotherapy in the head and neck area
* Severe hematologic disorders
* Any other diseases or medications that may compromise normal wound healing
* Pregnancy or nursing mother
* Contraindications and limitations of the MD as described in the instructions for use: during pregnancy or lactation, children, presence of acute infection in the surgical area, patients with known sensitivity to porcine material or collagen allergies.
* Vulnerable subjects
* Known or suspected non-compliance
* Drug or alcohol abuse
* Inability to follow the procedures of the investigation, e.g. due to language problems, psychological disorders, dementia, etc.
* Participation in another investigation with an investigational drug or another MD within the 30 days preceding and during the present investigation,
* Enrolment of the PI, his/her family members, employees and other dependent persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Volumetric dimensional changes | 0-5 years
  To assess the volumetric dimensional changes in pontic sites after site development using CTG compared to VCMX

SECONDARY OUTCOMES:
Clinical: PPD | 0-5 years
  Clinical: Probing depth in neighboring teeth
Clinical BoP | 0-5 years
  Clinical: Bleeding on probing
Clinical: Suppuration | 0-5 years
  Clinical: Suppuration on probing
Clinical: Mucosa | 0-5 years
  Clinical: Apical migration of the marginal mucosa
Clinical: ktw | 0-5 years
  Clinical: Keratinized tissue width
Clinical: Mobility | 0-5 years
  Clinical: Mobility
Clinical: Thickness | 0-5 years
  Clinical: Mucosal thickness
Clinical: Contributing factors | 0-5 years
  Clinical: Presence of local contributing factors
Patient-reported satisfaction | 0-5 years
  Questionnaire: Overall patient satisfaction with the treatment provided
Patient-reported esthetics | 0-5 years
  Questionnaire: Esthetics
Patient-reported discomfort | 0-5 years
  Questionnaire: Discomfort
Patient-reported pain | 0-5 years
  Questionnaire: Pain
Prosthetics Survival | 0-5 years
  Prosthetic-related: Fixed dental prostheses survival rates
Prosthetics Success | 0-5 years
  Prosthetic-related: Fixed dental prostheses success rates
Prosthetics Complications | 0-5 years
  Prosthetic-related: Technical complications
Prosthetics PES-WES | 0-5 years
  Prosthetic-related: Esthetic score (PES-WES)
Prosthetics: Occlusal | 0-5 years
  Prosthetic-related: Occlusal contacts (static and dynamic)
Prosthetics: Interproximal | 0-5 years
  Prosthetic-related: Presence of interproximal contacts.
Radiographics BL | 0-5 years
  Marginal bone levels
Radiographics PP | 0-5 years
  Periapical pathosis
Radiographics distance | 0-5 years
  Distance from the adjacent teeth/implants
Radiographics Contacts | 0-5 years
  Presence of open contacts

CONTACTS AND LOCATIONS:
Overall Officials: Manrique Fonseca, DDS, Principal Investigator — University of Bern
Locations (1):
- University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No